CLINICAL TRIAL: NCT04526106
Title: A First-in-Human Study of Highly Selective FGFR2 Inhibitor, RLY-4008, in Patients With Intrahepatic Cholangiocarcinoma (ICC) and Other Advanced Solid Tumors
Brief Title: REFOCUS: A First-in-Human Study of Highly Selective FGFR2 Inhibitor, RLY-4008, in Patients With ICC and Other Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Elevar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RLY-4008-101
Record Dates: First submitted 2020-08-07; First posted 2020-08-25 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: FGFR2 Amplification; FGFR2 Gene Mutation; FGFR2 Gene Fusion/Rearrangement; FGFR2 Gene Translocation; FGFR2 Gene Activation; Intrahepatic Cholangiocarcinoma; Cholangiocarcinoma; Other Solid Tumors, Adult
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Intervention Model Description: Part 1 (multiple ascending doses):
  • Unresectable or metastatic CCA or other unresectable or metastatic solid tumor
  Part 2 (RP2D determined in Part 1):
  * Group 1: CCA patients w/ an FGFR2 fusion previously treated w/ an FGFRi treatment
  * Group 2: CCA patients w/ an FGFR2 fusion w/ prior chemotherapy but no prior FGFRi treatment
  * Group 3: Non-CCA patients w/ an FGFR2 fusion and no prior FGFRi
  * Group 4: Non-CCA patients w/ an FGFR2 amplification and no prior FGFRi treatment
  * Group 5: Non-CCA patients w/ an FGFR2 mutation and no prior FGFRi treatment
  * Group 6: CCA patients w/ an FGFR2 fusion with no prior chemotherapy and no prior FGFRi treatment
  * Group 7: CCA patients w/ an FGFR2 mutation or amplification and no prior FGFRi treatment
  Part 3 (Extension of Part 2, Group 2):
  • CCA patients w/ an FGFR2 fusion with prior chemotherapy but no prior FGFRi treatment
  Part 4 (Rollover):
  • Ongoing Parts 1, 2, and 3 patients enrolled on study and receiving RLY-4008
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Dose Escalation (Experimental): Multiple doses of RLY-4008 for oral administration.
  Interventions: Drug: RLY-4008
- Part 2: Dose Expansion (Experimental): Oral dose of RLY-4008 as determined during Part 1 Dose Escalation.
  Interventions: Drug: RLY-4008
- Part 3: Extension (Experimental): Oral dose of RLY-4008 as determined during Part 1 Dose Escalation.
  Interventions: Drug: RLY-4008
- Part 4: Rollover (Experimental): Oral dose of RLY-4008 as determined during Part 1 Dose Escalation.
  Interventions: Drug: RLY-4008

INTERVENTIONS:
Drug: RLY-4008 — RLY-4008 is an oral inhibitor of FGFR2

SUMMARY:
This is a Phase 1/2, open-label, FIH study designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PDy), and antineoplastic activity of RLY-4008, a potent and highly selective FGFR2 inhibitor, in patients with unresectable or metastatic cholangiocarcinoma (CCA) and other solid tumors. The study consists of 4 parts: a dose escalation (Part 1), a dose expansion (Part 2), and an extension (Part 3) and a rollover (Part 4).

ELIGIBILITY:
Key Inclusion Criteria

* Histologically or cytologically confirmed unresectable or metastatic solid tumor
* Documented FGFR2 gene fusion, mutation, or amplification per local testing of blood and/or tumor
* Patient must have measurable disease per RECIST v1.1
* Patient has ECOG performance status of 0-1
* Patient must have disease that is refractory to standard therapy, disease that has not adequately responded to standard therapy, disease for which standard or curative therapy does not exist, or the patient must be intolerant to or have declined standard therapy
* Part 2 dose expansion patients with Cholangiocarcinoma:

  * Group 1: CCA patients with an FGFR2 fusion previously treated with an FGFRi
  * Group 2: CCA patients with an FGFR2 fusion with prior chemotherapy but not previously treated with an FGFRi
  * Group 6: CCA patients with an FGFR2 fusion with no prior chemotherapy and not previously treated with an FGFRi. Prior adjuvant/neo-adjuvant treatment completed >6 months before enrollment is acceptable. Up to 2 cycles of palliative chemotherapy are allowed during screening
  * Group 7: CCA patients with an FGFR2 mutation or amplification and not previously treated with an FGFRi. Note: For Group 7, patients with confirmed diagnosis of unresectable or metastatic CCA with an FGFR2 fusion are not eligible.
* Part 2 dose expansion patients with other solid tumors (NOT Cholangiocarcinoma):

  * Group 3: Non-CCA patients with an FGFR2 fusion and not previously treated with an FGFRi.
  * Group 4: Non-CCA patients with an FGFR2 amplification and not previously treated with an FGFRi.
  * Group 5: Non-CCA patients with an FGFR2 mutation and not previously treated with an FGFRi
* Part 3 extension:

  o CCA patients with an FGFR2 fusion with prior chemotherapy but not previously treated with an FGFRi
* Part 4:

  * Patient is receiving RLY-4008 on RLY-4008-101 study and benefiting from treatment as assessed by the investigator.

Key Exclusion Criteria

* Parts 1, 2, and 3

  * Ongoing, clinically significant FGFRi-induced retinal detachment or an ongoing clinically significant corneal or retinal disorder
  * Patient does not have adequate organ function (defined in protocol)
  * Patient has active infection, including human immunodeficiency virus (HIV), hepatitis B virus (HBV), and/or hepatitis C virus (HCV) (defined in protocol). Patients with well-controlled HBV are eligible (defined in protocol).
  * QT interval corrected using Fridericia's formula (QTcF) > 480 msec or history of prolonged QT syndrome, Torsades de pointes or familial history of prolonged QT syndrome
  * Clinically significant, uncontrolled cardiovascular disease
  * CNS metastases or primary CNS tumor that is associated with progressive neurologic symptoms
* Part 4:

  * Patient has permanently discontinued treatment with RLY-4008 for any reason before enrolling into Part 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2025-09-27 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Part 1 and Part 4: Number of patients with adverse events and serious adverse events | Every cycle (4-week cycles) until study discontinuation, approximately 24 months
Part 1: Determination of maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of RLY-4008 | Cycle 1 (4-week cycle) of treatment for MTD and at the end of every cycle (4-week cycles) for RP2D until study discontinuation, approximately 24 months
Part 2 and Part 3: Objective Response Rate (ORR) assessed by Independent Review Committee per RECIST v1.1 | Approximately every 8 weeks during treatment and every 12 weeks after the last dose in the absence of progressive disease, approximately 36 months
Part 4: Number of patients with dose interruptions | Every 28-day cycle until end of treatment, approximately 24 months.
Part 4: Number of patients with dose reductions | Every 28-day cycle until end of treatment, approximately 24 months.
Part 4: Number of patients with dose discontinuations | Every 28-day cycle until end of treatment, approximately 24 months.

SECONDARY OUTCOMES:
Part 1: FGFR2 gene status in plasma circulating tumor deoxyribonucleic acid (ctDNA) and tumor tissue | Every cycle (4-week cycles) through Cycle 3 and every other cycle thereafter until study discontinuation, approximately 24 months
Part 1: Duration of Response (DOR) assessed by Investigator per RECIST v1.1 | Approximately every 8 weeks during treatment and every 12 weeks after the last dose in the absence of progressive disease, approximately 36 months
Part 1: Disease Control Rate (DCR) as assessed by Investigator per RECIST v1.1 | Approximately every 8 weeks during treatment and every 12 weeks after the last dose in the absence of progressive disease, approximately 36 months
Part 1, Part 2, and Part 3: Objective Response Rate (ORR) as assessed by Investigator per RECIST v1.1 | Approximately every 8 weeks during treatment and every 12 weeks after the last dose in the absence of progressive disease, approximately 36 months
Pharmacokinetic parameters including maximum plasma drug concentration (Cmax) | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every cycle through Cycle 4 (4-week cycles)
Pharmacokinetic parameters including area under the plasma concentration versus time curve (AUC) | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every cycle through Cycle 4 (4-week cycles)
Pharmacokinetic parameters including half-life (t1/2) | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every cycle through Cycle 4 (4-week cycles)
Part 1: Pharmacodynamic parameters including changes in fibroblast growth factor 23 (FGF-23) | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every other cycle (4-week cycles) from Cycle 3, approximately 24 months
Part 1: Pharmacodynamic parameters including changes in carcinoembryonic antigen (CEA) | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every other cycle (4-week cycles) from Cycle 3, approximately 24 months
Part 1: Pharmacodynamic parameters including changes in cancer antigen 19-9 (CA 19-9) | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every other cycle (4-week cycles) from Cycle 3, approximately 24 months
Part 2 and Part 3: Duration of response (DOR) assessed by Investigator and Independent Review Committee per RECIST v1.1 | Approximately every 8 weeks during treatment and every 12 weeks after the last dose in the absence of progressive disease, approximately 36 months
Part 2 and Part 3: Progression-free survival (PFS) assessed by Investigator and Independent Review Committee per RECIST v1.1 | Approximately every 8 weeks during treatment and every 12 weeks after the last dose in the absence of progressive disease, approximately 36 months
Part 2 and Part 3: Disease control rate (DCR) assessed by Investigator and Independent Review Committee per RECIST v1.1 | Approximately every 8 weeks during treatment and every 12 weeks after the last dose in the absence of progressive disease, approximately 36 months
Part 2 and Part 3:Overall survival (OS) | Up to approximately 36 months.
Part 2 and Part 3:Change from baseline in quality of life as assessed by EORTC QLQ-C30 | Approximately every 4 weeks during treatment, approximately 24 months
Part 2 and Part 3:Dose intensity | Every 28-day cycle until end of treatment, approximately 24 months.
Part 2 and Part 3: Number of patients with dose interruptions | Every 28-day cycle until end of treatment, approximately 24 months.
Part 2 and Part 3: Number of patients with dose reductions | Every 28-day cycle until end of treatment, approximately 24 months.
Part 2 and Part 3: Number of patients with dose discontinuations | Every 28-day cycle until end of treatment, approximately 24 months.
Part 2 and Part 3: Correlation between FGFR2 genotype by central tissue assessment and antitumor response, as measured by ORR | Approximately every 8 weeks during treatment and every 12 weeks after the last dose in the absence of progressive disease, approximately 36 months

CONTACTS AND LOCATIONS:
Locations (48):
- United States (18):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic, Phoenix, Arizona
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Mayo Clinic, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Taussig Cancer Institute Cleveland Clinic, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Texas Oncology, Dallas, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - Virginia Mason Medical Center, Seattle, Washington
- Australia (3):
  - St. Vincent's Hosptial Sydney, Darlinghurst
  - Linear Clinical Research Ltd, Nedlands
  - Icon Cancer Care South Brisbane, South Brisbane
- France (4):
  - Institut Bergonie, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Centre Leon Berard, Lyon
  - Gustave Roussy Cancer Campus, Paris
- Germany (3):
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - LMU Klinikum, Campus Grosshadern, Munich
- Queen Mary Hospital, Hong Kong, Hong Kong
- Istituto Europeo di Oncologia, Milan, Italy
- Netherlands (2):
  - Netherlands Cancer institute, Amsterdam
  - Erasmus MC, Rotterdam
- National Cancer Center Singapore, Singapore, Singapore
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - START Barcelona-Hospital HM Nou Delfos, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Fundación Jiménez Díaz- START MADRID, Madrid
  - Hospital Universitario HM Sanchinarro-START MADRID-CIOCC, Madrid
  - Clinica de Universidad de Navarra, Pamplona
  - Hospital Clínico Universitario de Valencia, Valencia
- Karolinska University Hospital, Stockholm, Sweden
- China Medical University Hospital, Taichung, Taiwan
- United Kingdom (4):
  - Guy's Hospital, London
  - Sarah Cannon Research Institute UK, London
  - University College London Hospitals NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No